CLINICAL TRIAL: NCT07007728
Title: Efficacy and Safety of Iparomlimab/Tuvonralimab Combined With Bevacizumab and CAPEOX as Conversion Therapy in Patients With Right-Sided or RAS-mutant, Microsatellite Stable, Initially Unresectable Colorectal Cancer Liver Metastasis: A Prospective, Open-Label, Single-Arm, Single-Center, Phase II Clinical Trial
Brief Title: Iparomlimab/Tuvonralimab Combined With Bevacizumab and CAPEOX as Conversion Therapy for Colorectal Cancer Liver Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wang Kun, MD, Prof, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DUALTRANSFORM (PKUCRLM-02)
Record Dates: First submitted 2025-05-15; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Neoplasms; Secondary Malignant Neoplasm of Liver
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab/Tuvonralimab Combined with Bevacizumab and CAPEOX (Experimental)
  Interventions: Drug: Iparomlimab/Tuvonralimab; Drug: Bevacizumab + CAPEOX; Procedure: Surgical resection ± ablation or stereotactic radiotherapy (if applicable)

INTERVENTIONS:
Drug: Iparomlimab/Tuvonralimab — 5mg/kg intravenous infusion on Day 1 of each cycle (every 21 days). Duration: 3 or 6 cycles
Drug: Bevacizumab + CAPEOX — Bevacizumab: 7.5mg/kg intravenous infusion on Day 1 of each cycle (every 21 days).
  Capecitabine: 1000 mg/m2 twice daily orally on Day 1-14 of each cycle (every 21 days).
  Oxaliplatin: 130 mg/m2 intravenous infusion on Day 1 of each cycle (every 21 days).
  Duration:
  Conversion therapy phase: 3 or 6 cycles; Postoperative follow-up phase (for patients with successful conversion surgery ): 3 or 6 cycles (a total perioperative duration of 9 cycles); Maintenance phase (for patients without successful conversion surgery ): Continuous therapy until disease progression, intolerable adverse events, withdrawal of consent, loss to follow-up, death, or study termination.
Procedure: Surgical resection ± ablation or stereotactic radiotherapy (if applicable) — After 3 or 6 cycles of conversion therapy, surgical resection ± ablation or stereotactic radiotherapy will be provided if applicable.

SUMMARY:
More than half of colorectal cancer (CRC) patients present with RAS mutations or right-sided primary tumors; however, objective response rates (ORRs) to bevacizumab combined with chemotherapy remain suboptimal. Additionally, approximately 95% of metastatic CRC (mCRC) cases are microsatellite stable (MSS), where immune checkpoint inhibitor monotherapy demonstrates limited efficacy, necessitating combination strategies. Iparomlimab/tuvonralimab is the first bifunctional combination of anti-PD-1/anti-CTLA-4 monoclonal antibodies, which has shown therapeutic promise in first-line mCRC when combined with bevacizumab and capecitabine plus oxaliplatin (CAPEOX). Nevertheless, whether improved treatment response rates in mCRC patients can lead to higher surgical conversion rates remains unclear. This study evaluates the efficacy and safety of iparomlimab/tuvonralimab combined with bevacizumab and CAPEOX as conversion therapy in patients with right-sided or RAS-mutant, MSS, initially unresectable colorectal cancer liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria will be included in this study:

1. Sign written informed consent before initiating any trial-related procedures;
2. ≥18 years and ≤79 years old, regardless of gender;
3. Pathologically confirmed colorectal adenocarcinoma with liver metastases confirmed by pathology or imaging;
4. No prior first-line systemic therapy (e.g., targeted therapy, immunotherapy, systemic chemotherapy) for liver metastases;
5. At least one radiographically measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST version 1.1);
6. Multidisciplinary team (MDT)-confirmed initially unresectable liver metastases (criteria for unresectability: inability to achieve R0/R1 resection via surgery, or anticipated residual liver volume <30% post-resection, or inability to preserve adequate hepatic inflow/outflow for residual liver). Patients with extrahepatic metastases (excluding brain/bone metastases) amenable to local treatment are eligible;
7. Genetic testing results confirming either RAS mutation or right-sided colon location with RAS wild-type status, absence of BRAF V600E mutation, and microsatellite stability (MSS)/proficient mismatch repair (pMMR) confirmed through immunohistochemistry (IHC) or PCR testing.
8. ECOG performance status score 0-1;
9. Life expectancy ≥12 weeks;
10. No indications for emergency surgery due to primary tumor complications including significant bleeding or obstruction;
11. Adequate organ function meeting the following laboratory parameters:

    i. Absolute neutrophil count (ANC) ≥1.5×10^9/L without granulocyte colony-stimulating factor support within 14 days; ii. Platelet count (PLT) ≥75×10^9/L without transfusion within 14 days; iii. Hemoglobin (HGB) >70 g/L without transfusion or erythropoietin use within 14 days; iv. Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); serum albumin (Alb) ≥28.0 g/L; v. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5×ULN; vi. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 mL/min; vii. Normal coagulation function: International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5×ULN;
12. Fertile female patients or male patients with fertile partners must agree to use highly effective contraception (failure rate <1% per year) from 7 days before first dose until 24 weeks post-treatment;
13. Fertile female patients must have negative serum pregnancy test within 7 days before first dose;
14. Patients must be capable of and willing to comply with study protocol requirements, including scheduled visits, treatment plans, laboratory tests, and other trial-related procedures.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will be excluded from this study:

1. Patients intolerant to systemic chemotherapy or surgery;
2. Liver metastases occurring during or within 6 months after oxaliplatin-based adjuvant chemotherapy for the primary tumor;
3. Major surgery within 6 weeks before treatment initiation, anticipated requirement for major surgery during the study, or presence of severe traumatic injury, fractures, ulcers, or non-healing wounds;
4. History of myocardial infarction, severe/unstable angina, coronary artery bypass grafting, or heart failure (NYHA class III-IV) within 3 months before treatment initiation;
5. Prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1/L1, CTLA-4 inhibitors);
6. Concurrent or prior malignancies;
7. History of autoimmune diseases or allogeneic stem cell/solid organ transplant (excluding corneal transplant) rendering immunotherapy intolerance;
8. Moderate-to-severe allergic reactions, hypersensitivity, or intolerance to antibody-based therapies;
9. Clinically significant bleeding symptoms or high bleeding risk within 3 months before treatment initiation (e.g., gastrointestinal bleeding, gastroesophageal varices, hemorrhagic gastric ulcer, or history of hematochezia, hematemesis, or hemoptysis);
10. Clinically symptomatic ascites/pleural/pericardial effusion requiring therapeutic intervention;
11. Primary tumor obstruction, perforation or intra-abdominal infection within 3 months before treatment initiation, without appropriate management;
12. Known hypersensitivity to active pharmaceutical ingredient or excipients of the investigational drug;
13. Dysphagia, active peptic ulcer, intestinal obstruction, active gastrointestinal bleeding, gastrointestinal perforation, malabsorption syndrome, or uncontrolled inflammatory bowel disease;
14. Pregnant or breastfeeding women;
15. Concurrent participation in other clinical trials;
16. Any other condition deemed inappropriate for study participation by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Following 3 or 6 cycles (each cycle is ~21 days) of the treatment, approximately 9 or 18 weeks overall
  The proportion of subjects achieving complete response or partial response, assessed by investigators according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Surgical Conversion Rate | Following 3 or 6 cycles (each cycle is ~21 days) of the treatment, approximately 9 or 18 weeks overall
  The proportion of subjects with successful conversion surgery. The criteria for successful conversion are as follows: evaluation of liver metastases achieves partial response after the conversion therapy; liver tumor-free status can be achieved through surgical resection ± ablation or stereotactic radiotherapy, with a residual liver volume exceeding 40%; liver function is classified as Child-Pugh Class A, and other liver function and laboratory parameters meet surgical and anesthesia requirements.
Major Pathological Response Rate | Perioperative/Periprocedural
  The proportion of subjects in whom postoperative pathological evaluation of liver metastases shows either no residual tumor cells (complete regression) or residual tumor cells comprising 1-49% of the specimen.
Progression-free Survival | From the date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  The time from the initiation of treatment until disease progression or death from any cause, whichever occurs first.
Overall Survival | From the date of treatment initiation until the date of death from any cause, assessed up to 18 months
  The time from the initiation of treatment until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The investigator has no individual patient data (IPD) sharing plan.